Official Title: The effects of spasticity on glucose metabolism and soft tissue body composition in individuals with motor complete and motor incomplete spinal cord injury

NCT03859960

Document date: August 6th, 2020

## Statistical analysis

The IBM SPSS Statistics 22 (IBM SPSS, Turkey) program was used for the statistical analysis. Normal distribution was evaluated using the Shapiro-Wilk test. Descriptive statistics of mean, SD, and frequencies were calculated. Pearson correlation analysis was used to assess the association between the parameters with conformity to the normal distribution. Statistical significance was evaluated at p<0.05.